CLINICAL TRIAL: NCT06946342
Title: "Efficacy of the WATERinMOTION Aquatic Exercise Program Compared to Land-Based Rehabilitation on Low-Back Pain Relief and Quality of Life in Sedentary Overweight and Obese Middle-Aged Women: A Randomized Controlled Trial"
Brief Title: WATERinMOTION Aquatic Exercise Program Compared to Land-Based Rehabilitation on Low-Back Pain Relief and Quality of Life
Acronym: WATERinMOTION
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sistan and Baluchestan (Other)
Responsible Party: Principal Investigator, Mohammadreza Rezaeipour, Assoc.Prof.Dr, University of Sistan and Baluchestan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9378-30 - 1 - 2025; 9378 (Registry Identifier: Ferdows Shafa)
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Low Back Pain; Obesity; Sedentary Behavior
Keywords: Hydrotherapy; Exercise Therapy; Middle Aged; Quality of Life; Disability Evaluation
MeSH Terms: conditions — Low Back Pain; Obesity; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: This is a two-arm, randomized, single-blind, parallel-group trial comparing the efficacy of two distinct exercise interventions:
  Experimental Arm: Structured aquatic exercise program (WATERinMOTION).
  Active Comparator Arm: Land-based rehabilitation program.
Who Masked: Outcomes Assessor
Masking Description: Single-blind (outcome assessors only; participants/instructors unblinded due to intervention nature).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Aquatic Exercise Group (Experimental): "60-minute WATERinMOTION sessions (3x/week for 8 weeks) in a heated pool (30-32°C), including aerobic, strength, and flexibility exercises."
  Interventions: Behavioral: "Aquatic Exercise Group"
- "Land-Based Rehabilitation Group" (Active Comparator): "60-minute land-based sessions (3x/week for 8 weeks), including core stabilization, low-impact aerobics, and stretching."
  Interventions: Behavioral: Land-Based Rehabilitation Group"

INTERVENTIONS:
Behavioral: "Aquatic Exercise Group" — "Structured WATERinMOTION aquatic exercise program (3x/week for 8 weeks) in a heated pool (30-32°C), including warm-up, aerobic conditioning, resistance training with water equipment (e.g., dumbbells, noodles), and cool-down. Sessions are group-based and led by certified instructors."
  Arms: "Aquatic Exercise Group
Behavioral: Land-Based Rehabilitation Group" — "60-minute land-based sessions (3x/week for 8 weeks), including core stabilization, low-impact aerobics, and stretching."
  Arms: "Land-Based Rehabilitation Group"

SUMMARY:
This randomized controlled trial compares the efficacy of an 8-week WATERinMOTION aquatic exercise program versus land-based rehabilitation for reducing low-back pain (LBP) and improving quality of life in sedentary, overweight/obese middle-aged women (n=45). Outcomes include pain intensity (VAS), functional disability (ODI), and health-related quality of life (SF-36).

DETAILED DESCRIPTION:
Participants (aged 45-65, BMI ≥25 kg/m², chronic LBP ≥3 months) were randomized to aquatic exercise (n=45) or land-based rehabilitation (n=45). Both groups completed three 60-minute sessions/week for 8 weeks. Assessments occurred at baseline, post-intervention, and 3-month follow-up. Primary outcomes: VAS and ODI; secondary outcomes: SF-36 and satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 45-65, BMI ≥25 kg/m².
* Sedentary (<150 min/week moderate activity).
* Chronic LBP (≥3 months, VAS ≥4).

Exclusion Criteria:

* Contraindications to exercise (e.g., severe cardiovascular disease).
* Spinal surgery history or inflammatory conditions (e.g., rheumatoid arthritis).

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Baseline, 8 weeks (post-intervention), 3-month follow-up
  Visual Analog Scale (VAS), Scale Range: 0 (no pain) to 10 (worst pain imaginable),
Functional Disability | Baseline, 8 weeks (post-intervention), 3-month follow-up
  Oswestry Disability Index (ODI), Scale Range: 0% (no disability) to 100% (severe disability)

SECONDARY OUTCOMES:
Health-Related Quality of Life (HRQoL) | Baseline, 8 weeks (post-intervention), 3-month follow-up
  Measure: 36-Item Short Form Survey (SF-36)
Participant Satisfaction | 8 weeks (post-intervention), 3-month follow-up
  Measure: 5-point Likert Scale, Scale Range: 1 (very dissatisfied) to 5 (very satisfied)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammadreza Rezaeipour, MD, PhD, Study Director — Assoc.Prof.Dr. of University of Sistan and Baluchestan, Zahedan, Iran
Locations (1):
- Sport Sciences Department, Zahedan, Sistan and Baluchestan, Iran

IPD SHARING:
Plan to Share IPD: No
Privacy concerns (sensitive health data of overweight/obese women/men).
  Lack of pre-specified data-sharing plan in ethics approval.